CLINICAL TRIAL: NCT04869449
Title: Neuro-pharmacological Properties of Repurposed Ketoconazole in Glioblastomas: A Phase 0 Clinical Trial
Brief Title: Neuro-pharmacological Properties of Repurposed Ketoconazole in Glioblastomas
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrollment was stopped due to direction from the scientific review committee of the Penn State Cancer Institute. The instruction came due to slow accrual.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Alireza Mansouri, Assistant Professor, Department of Neurosurgery, Penn State Health Milton S Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00014115
Record Dates: First submitted 2021-04-13; First posted 2021-05-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioblastoma Multiforme of Brain; Glioblastoma Multiforme, Adult
Keywords: Glioblastoma; Glioblastoma Multiforme; GBM; Brain cancer; Ketoconazole; Anti-fungal agents
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketoconazole (Experimental): Participants will be taking 400 mg of the study drug (two 200 mg tablets) by mouth twice a day until the day of biopsy or surgery. On the day of biopsy or surgery, participants will take their medication the morning of their biopsy or surgery (before the operation) and in the evening after their biopsy or surgery (after the operation). Participants will then take the last dose of the medication in the morning of the day after their biopsy or surgery. Participants will be given 12 days' worth of the study drug (pills) and verbally instructed how and when to take them.
  Interventions: Drug: Ketoconazole

INTERVENTIONS:
Drug: Ketoconazole — 400 mg (two 200 mg tablets) orally
  Other Names: Nizoral

SUMMARY:
This research is being done to find out if the study drug (ketoconazole) can enter brain tumors at a high enough amount to stop the tumor cells from dividing. Ketoconazole is a drug which doctors already use for fungal infections and is thought to be able to effect tumor cells. As treatments for this type of brain tumor are limited, it is hoped that the results of this study will help to determine if the study drug should be studied further as a possible treatment.

DETAILED DESCRIPTION:
Both ketoconazole and posaconazole are FDA-approved anti-fungal agents with a well-established side effect and safety profile. Ketoconazole and posaconazole have shown efficacy in reducing tumor cell proliferation in in-vitro studies. Furthermore, both have also shown efficacy, mediated at least in part through inhibition of hexokinase 2 (HK2) activity, in animal models with dosing concentration and schedules that are documented as safe in humans. As a drug, posaconazole has a more predictable half-life than ketoconazole and has less off-target effects. Therefore, the proposed trial will focus on the role of posaconazole exclusively. As a first step, demonstration of adequate penetrance of study drug in brain and tumor tissue (pharmacokinetics) and biological effect (inhibition of glycolysis and subsequent tumor cell death) is necessary prior to large scale clinical studies. A total of 5 control participants will be included in this study as the investigator specifically wants to assess for pharmacodynamic differences too. The addition of a control group to this study rather to both the studies (ketoconazole study is a separate protocol) is because the investigator feels posaconazole may be a more promising drug for moving forward.

Plasma drug concentration measurements are an unreliable method to assess delivery of drugs across the blood-brain barrier. In contrast, intracerebral microdialysis catheters (MDC) monitoring allows for approximate measurements within extracellular fluid (ECF) sampling of the brain. MDC placement within the brain is not a novel technique and has been utilized routinely in the ICU setting to measure brain metabolism by sampling of ECF of traumatic brain injury patients.

MDC are now FDA-approved and are being placed routinely with intracranial pressure monitors. This method allows for continuous measurement of ECF within a tumor or normal tissue. The dialysis probe has a semipermeable membrane which is less than 1 mm in diameter into which two sections of microcatheter are fused. Previous studies have demonstrated the feasibility of keeping the catheters in place of critically injured patients for up to 2 weeks.

When placed at the time of surgical resection, the microcatheters are stereotactically implanted, placing the probe within the desired brain and/or tumor region. Externally, the catheter is connected to a syringe pump, which delivers a low flow rate (μl/min) of continuous perfusion fluid (Lactated Ringers or artificial CSF) and dialysate is collected in a microvial from the outlet tube. This sterile, single use catheter is minimally invasive and developed to achieve optimal diffusing characteristics similar to passive diffusion of a capillary blood vessel. Just as in the function of brain capillary vessel, water, inorganic ions and small organic molecules freely diffuse across the membrane of the probe, whereas proteins and protein bound compounds are impermeable. Additionally, lipophilic compounds are poorly recovered. Therefore, assessment of pharmacokinetics of drug using MDC provides valuable insight relevant to its anti-neoplastic properties.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Evidence of primary or recurrent high-grade gliomas (HGG) that in the opinion of the treating team would require surgical resection
* Karnofsky Performance Score (KPS) ≥ 60%
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy greater than 12 weeks
* Adequate liver function defined as Alanine aminotransferase (ALT),Aspartate transaminase (AST), Alkaline phosphatase (ALP) within 1.5x institutional upper limit of normal
* Adequate renal function defined as estimated glomerular filtration rate (eGFR) levels within 1.5x the institutional upper limit of normal
* Ability to swallow medication
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation.
* Ability to understand and willingness to sign a written informed consent document
* Be able to comply with treatment plan, study procedures and follow-up examinations

Exclusion Criteria:

* Patients may not be receiving any other investigational agents while on study
* Patients who have known allergy to ketoconazole or other azoles
* Patients who have previously had a severe side effect, such as agranulocytosis and neutropenia, in conjunction with previous azole class drugs for a parasitic infection
* Patients with a history of acute or chronic hepatitis
* Patients with liver enzymes (ALT, AST, ALP) >1.5x above normal range for the laboratory performing the test
* Patients who are taking metronidazole and cannot be safely moved to a different antibiotic greater than 7 days prior to starting ketoconazole therapy
* Patients who are taking any anti-convulsant medication that interferes with the cytochrome P450 pathway (e.g. phenytoin, phenobarbital, carbamazepine, etc.) and who cannot be switched to alternative medications such as keppra (levetiracetam)
* Uncontrolled intercurrent illness such as chronic hepatitis, acute hepatitis, or psychiatric illness/social situation that would limit compliance with study requirements
* Patients with a history of Addison's disease or other forms of adrenal insufficiency
* Patient with little or no stomach acid production (achlorhydria)
* Pregnant and breast feeding women
* Patients with a history of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product administration or may interfere with the interpretation of the results.
* Patients who are not available for follow-up assessments or unable to comply with study requirements.
* Patients who are currently taking medications that induce the metabolism of ketoconazole, such as isoniazid, nevirapine, rifamycins (such as rifabutin, rifampin), or St. John's wort and cannot be safely discontinued off of them for the duration of the trial.
* Patients who are currently taking medications for which the metabolism may be affected by ketoconazole, which include but are not limited to: benzodiazepines (such as alprazolam, midazolam, triazolam), domperidone, eletriptan, eplerenone, ergot drugs (such as ergotamine), nisoldipine, drugs used to treat erectile dysfunction (ED) or pulmonary hypertension (such as sildenafil, tadalafil), some drugs used to treat seizures (such as carbamazepine, phenytoin), some statin drugs (such as atorvastatin, lovastatin, simvastatin).
* Patients who are non-English speakers
* Patients who are not capable of understanding the consent form and would need a legally authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Establish drug concentration versus time profile yielding maximum plasma concentration (Cmax) | Collected over a 24-hour period after surgery (biopsy or resection)
  Assessment of the concentration versus time curves of drug in the dialysate fluid
Establish drug concentration versus time profile yielding half-life pharmacodynamics | Collected over a 24-hour period after surgery (biopsy or resection)
  Assessment of the concentration versus time curves of drug in the dialysate fluid

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events as assessed by CTCAE v 5.0 | from Baseline to Visit 7 (14 days +/- 7 days post-op)
  Measured through the Grade and Frequency of adverse events, based on the CTCAE v5.0 criteria
Hexokinase activity assay- measured as a proportion of hexokinase enzyme activity in relation to positive control | Within 24 hours after tumor resection
  Measured using a hexokinase assay on tumor tissue
Concentration of lactate measured using mass spectrometry in resected tumor tissue | Immediately after biopsy or resection of tissue
  Measured using mass spectrometry
Concentration of pyruvate, measured using mass spectrometry in resected tumor tissue | Immediately after biopsy or resection of tissue
  Measured using mass spectrometry
Evaluate ketoconazole's effect on tumor proliferation in tumor tissue | Within 24 hours after biopsy or tumor resection
  Measured using Ki-67 proliferation index
Evaluate ketoconazole's effect on cell death in tumor tissue | Within 24 hours after biopsy or tumor resection
  Measured using TUNEL staining
Evaluate ketoconazole's effect on angiogenesis in tumor tissue | Within 24 hours after biopsy or tumor resection
  Based on expression of vascular endothelial growth factor (VEGF)
Correlation of concentration versus time profile of ketoconazole , compared to that of lactate - measured using mass spectrometry over 24 hours | Over the same 24-hour period used to measure the concentration of drug
  Assessed based on the concentration versus time profile of lactate in the dialysate fluid
Correlation of concentration versus time profile of ketoconazole, compared to that of pyruvate - measured using mass spectrometry over 24 hours | Over the same 24-hour period used to measure the concentration of drug
  Assessed based on the concentration versus time profile of pyruvate in the dialysate fluid

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Mansouri, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No